CLINICAL TRIAL: NCT00233389
Title: A Post-marketing Clinical Study of Rebamipide to Investigate the Gastric Ulcer Healing Effect of Continued Dosing Following Helicobacter Pylori Eradication Therapy
Brief Title: Post-marketing Clinical Study of Rebamipide in Patients With Gastric Ulcer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C03700-003; JapicCTI-050035
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Stomach Ulcer
MeSH Terms: conditions — Stomach Ulcer | interventions — rebamipide

INTERVENTIONS:
Drug: Rebamipide

SUMMARY:
To examine the efficacy of continued administration of rebamipide following bacteria eradication therapy in patients with H. pylori-positive active gastric ulcer in a placebo-controlled, double-blind study

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 years or older at time of consent
2. H. pylori-positive patients meeting both of the following criteria:• Assessed as H. pylori-positive by rapid urease test and/or 13C-urea breath test at pre-study examination, • Assessed as H. pylori-antibody-positive by urine-based test after obtaining informed consent
3. Patients endoscopically diagnosed with gastric ulcer meeting the following criteria:• Active (A1- or A2-stage by Sakita/Miwa classification）, • Solitary, • Longitudinal diameter: ->5 mm
4. Patients who have not received proton pump inhibitors (PPIs), antibacterial agents, or antiprotozoal agents within 1 week prior to endoscopy

Exclusion Criteria:

1. Patients who have previously received H. pylori eradication therapy
2. Patients with acute gastric ulcer
3. Patients with linear ulcer
4. Patients with complication of duodenal ulcer (excluding cicatrix)
5. Patients who have undergone upper-GI tract or vagal nerve resection
6. Patients who are unsuitable for pharmacotherapy, e.g., with perforation or pyloric stenosis
7. Patients with gastric ulcer considered likely to induce massive hemorrhage (e.g., with obviously exposed blood vessels at lesion sites)
8. Patients with a history of amoxicillin shock
9. Patients with infectious mononucleosis
10. Patients with severe renal disorders
11. Patients with a history of hypersensitivity to penicillins, clarithromycin, lansoprazole, or rebamipide
12. Patients who have been treated with drugs contraindicated to clarithromycin, such as terfenadine, cisapride, and pimozide
13. Patients who are pregnant, possibly pregnant, lactating, or who desire to become pregnant during the study
14. Patients who are otherwise judged inappropriate for inclusion in the study by the investigator or subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2004-04-30 (Actual); Primary Completion 2005-09-01 (Actual); Study Completion 2005-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Division of New Product Evaluation and Development
Locations (1):
- Otsuka Pharmaceutical Co., Ltd., Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following the eradication therapy period, 154 subjects in the rebamipide group and 147 subjects in the placebo group, excluding withdrawals during the eradication therapy period, received the investigational medicinal product (IMP) (rebamipide or placebo) for the treatment of gastric ulcer.
Groups:
- Rebamipide: Following 1 week of H. pylori eradication therapy, a rebamipide 100 mg tablet was administered orally three times a day for 7 weeks.
- Placebo: Following 1 week of H. pylori eradication therapy, a placebo tablet was administered orally three times a day for 7 weeks.
Period: Overall Study
Arm/Group | Rebamipide | Placebo
Started | 154 | 147
Completed | 136 | 131
Not Completed | 18 | 16
Not completed — Adverse Event | 5 | 5
Not completed — Lack of Efficacy | 11 | 8
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Efficacy Analysis Set: Subjects who received H. pylori eradication therapy as specified and at least one dose of the IMP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rebamipide | Placebo | Total
Number analyzed (Participants) | 154 | 147 | 301
Age, Customized [Count of Participants; unit: Participants]
  20-39 years | 21 | 19 | 40
  40-59 years | 99 | 84 | 183
  >=60 years | 34 | 44 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 48 | 100
  Male | 102 | 99 | 201
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 154 | 147 | 301

OUTCOME MEASURES:

1. Primary Outcome: Gastric Ulcer Healing Rate (Number of Subjects Whose Gastric Ulcer Was Healed/Number of Subjects Evaluated x 100) at Week 8
Description: The percentage of subjects in the analysis set in whom endoscopic assessment of gastric ulcer stage (Sakita-Miwa Classification: A1, A2, H1, H2, S1, or S2) at 8 weeks after trial treatment (H. pylori eradication therapy + IMP) was judged as healed (S1 or S2) was calculated and evaluated by group.
Time Frame: Week 8
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rebamipide | Placebo
Number analyzed (Participants) | 154 | 147
percentage of participants | 70.13 [62.90 to 77.36] | 60.54 [52.64 to 68.45]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the start of IMP administration to 7 weeks or withdrawal.
Description: Safety analysis set included all subjects who received the IMP at least once and from whom data on at least 1 safety endpoint were obtained after the start of IMP.
Arm/Group | Rebamipide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/147
Serious Adverse Events (participants affected / at risk) | 2/154 | 1/147
Other Adverse Events (participants affected / at risk) | 85/154 | 75/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebamipide (N=154) | Placebo (N=147)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebamipide (N=154) | Placebo (N=147)
Cheilitis (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 27 | 27
Faeces hard (Gastrointestinal disorders) | 1 | 2
Gastric ulcer (Gastrointestinal disorders) | 5 | 2
Glossitis (Gastrointestinal disorders) | 0 | 3
Reflux oesophagitis (Gastrointestinal disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 16 | 15
Joint sprain (Injury, poisoning and procedural complications) | 2 | 0
Blood urea increased (Investigations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 3 | 1
White blood cell count decreased (Investigations) | 2 | 1
White blood cell count increased (Investigations) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 14 | 11
Headache (Nervous system disorders) | 7 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No